CLINICAL TRIAL: NCT03150602
Title: A Multi-Center, Open-Labelled, Pralatrexate Study in Asian Patients With Peripheral T-cell Lymphoma After Prior Therapy
Brief Title: A Pralatrexate Study in Asian Patients With Peripheral T-cell Lymphoma After Prior Therapy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taiwan Mundipharma Pharmaceuticals Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FOT14-TW-401
Record Dates: First submitted 2017-05-05; First posted 2017-05-12 (Actual); Last update posted 2017-05-12 (Actual); Status verified 2017-05

CONDITIONS: Peripheral T Cell Lymphoma; Progression, Disease
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral; Disease Progression | interventions — 10-propargyl-10-deazaaminopterin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pralatrexate treatment (Experimental): Pralatrexate will initially be administered at a dose of 30 mg/m2/week on days 1, 8, 15, 22, 29 and 36 for 6 weeks in a 7-week cycle (cycle: 6 weeks + 1 week rest). The scheduled date can be done within a window time of plus or minus 1 day
  Interventions: Drug: Pralatrexate

INTERVENTIONS:
Drug: Pralatrexate — This is a single arm study. Pralatrexate will be administered via IV over 3-5 minutes into a IV line containing normal saline (0.9% sodium chloride, NaCl) with the initial dose of 30 mg/m2/week on days 1, 8, 15, 22, 29, and 36 for 6 weeks in a 7-week cycle. The scheduled date can be done within a window time of plus or minus 1 day. The pralatrexate dose may be reduced to 20 mg/m2/week or omit if a patient experiences adverse events. Pralatrexate administration can be up to 5 cycles or until subject meets withdrawal criteria.
  Other Names: Folotyn

SUMMARY:
This study is to evaluate the objective response rate to pralatrexate in Asian PTCL patients after prior treatment failure, as determined by independent imaging reviewer(s) using international workshop lymphoma response criteria (IWC)

DETAILED DESCRIPTION:
Peripheral T-cell lymphomas (PTCL) are a group of aggressive and diverse lymphoproliferative disorders. It is characterized by the presence of malignant mature T-cells or NK cells. There is as yet no consensus regarding standard frontline or relapsed/refractory therapy for PTCL.

A previous phase II study conducted in US showed durable responses of pralatrexate treatment in relapsed or refractory PTCL, irrespective of age, histological subtypes, amount of prior therapy, prior methotrexate, and prior autologous stem-cell transplant. This single-arm, multi-center study aims to evaluate the efficacy and safety of pralatrexate monotherapy in prior treatment failure PTCL patients who may undergo HSCT in case of CR or PR, or continue pralatrexate in case of CR, PR or SD.

Primary objective:

* To evaluate the objective response rate to pralatrexate in Asian PTCL patients after prior treatment failure, as determined by independent imaging reviewer(s) using international workshop lymphoma response criteria (IWC)

Secondary objectives:

* To determine the safety of pralatrexate in Asian PTCL patients by,

  * Incidence of adverse events (AEs) and serious adverse events (SAEs) emergent from the treatment
* To evaluate the efficacy of pralatrexate in Asian PTCL patients after prior treatment failure by,

  * Overall survival (OS), progression-free-survival (PFS), complete response (CR) and partial response (PR) rate, and duration of CR and PR
  * Treatment duration with pralatrexate in the patients without hematopoietic stem cell transplant (HSCT) who achieve CR or PR
  * Percentage of patients who undergo HSCT
  * 1-year OS, 1-year PFS, and 1-year relapse rate after HSCT
  * 2-year OS, 2-year PFS, and 2-year relapse rate after HSCT

ELIGIBILITY:
Inclusion Criteria:

1. At least 20 years of age, inclusive
2. Patients with histologically/cytologically confirmed PTCL using either: NCCN diagnosis criteria, the Revised European American Lymphoma (REAL), and World Health Organization (WHO) disease classification (PTCL histology/cytology subtypes diagnosed by site investigators, PTCL histology/cytology subtypes rechecked by study central pathology lab):

   1. At least 5 patients with Peripheral T-cell lymphoma, NOS
   2. At least 5 patients with Angioimmunoblastic T-cell lymphoma
   3. At least 5 patients with Extranodal NK/T-cell lymphoma, nasal type
   4. Enteropathy-type T-cell lymphoma
   5. Hepatosplenic T-cell lymphoma
   6. Subcutaneous panniculitis-like T-cell lymphoma
   7. Adult T-cell lymphoma/leukemia (human T-cell leukemia virus [HTLV] 1+)
3. Patients with documented progressive disease (PD) failed after prior treatment

   1. Patients may not have received an experimental drug as their only prior therapy
   2. Patient has had at least 1 biopsy from initial diagnosis of PTCL or in the relapsed setting to confirm PTCL subtypes
   3. Patient has recovered from the toxic effects of prior therapy
4. Eastern Cooperative Oncology Group (ECOG) Performance Status ≤ 2.
5. Adequate hematological, hepatic, and renal function as defined by: absolute neutrophil count (ANC) ≥ 1000/µL, platelet count ≥ 100,000/µL (and ≥ 50,000/µL for any following dose), total bilirubin ≤ 1.5 mg/dL, aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 X upper limit of normal (ULN) (AST/ALT < 5 X ULN if documented hepatic involvement with lymphoma), creatinine ≤ 1.5 mg/dL or a calculated creatinine clearance ≥ 50 mL/min.
6. Women of childbearing potential must agree to practice medically acceptable contraceptive regimen from 30 days prior to study treatment initiation until at least 30 days after the last administration of pralatrexate and must have had a negative serum pregnancy test within 14 days prior to the first day of study treatment. Patients who are postmenopausal for at least 1 year (> 12 months since last menses) or were surgically sterilized do not require this test.
7. Men who are not surgically sterile must agree to practice a medically acceptable contraceptive regimen from study treatment initiation until at least 90 days after the last administration of pralatrexate.
8. Patient has provided written informed consent (IC)

Exclusion Criteria:

1. Patient has following subtypes (histologically/cytologically confirmed) of PTCL

   1. Anaplastic large cell lymphoma, ALK +/-
   2. Patient has: Precursor T/NK neoplasms, with the exception of blastic NK lymphoma
   3. T-cell prolymphocytic leukemia (T-PLL)
   4. T-cell large granular lymphocytic leukemia
   5. Mycosis fungoides and transformed mycosis fungoides
   6. Sézary syndrome
   7. Primary cutaneous CD30+ disorders: Anaplastic large cell lymphoma and lymphomatoid papulosis
   8. Patient has: Extranodal NK/T-cell lymphoma, nasal type with local recurrence
2. Active concurrent malignancy (except for non-melanoma skin cancer or carcinoma in situ of the cervix). If there is a history of prior malignancy, the patient must be disease-free for ≥ 5 years.
3. Congestive heart failure Class III/IV according to the New York Heart Association's Heart Failure guidelines.
4. Patients with human immunodeficiency virus (HIV)-positive diagnosis and are receiving combination anti-retroviral therapy.
5. Current or the history of brain metastases or central nervous system (CNS) diseases
6. Have undergone allogeneic stem cell transplant
7. Relapsed less than 75 days from time of autologous stem cell transplant
8. Patients with uncontrolled hypertension, active uncontrolled infection, underlying medical condition including unstable cardiac disease, or other serious illness that would impair the ability of the patient to receive protocol treatment
9. Had major surgery within 2 weeks of study entry
10. Receipt of any conventional chemotherapy or radiation therapy (RT) within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to study treatment or planned use during the course of the study
11. Receipt of corticosteroids within 7 days of study treatment, unless patient has been taking a stable dose of no more than 10 mg/day of prednisone for at least 1 month
12. Use of any investigational drug, biologic modifier, or device within 4 weeks prior to study treatment or planned use during the course of the study
13. Previous exposure to pralatrexate
14. Other conditions that investigators consider not suitable for study enrollment

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2016-08-30 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | Up to 35 weeks
  Objective response rate (ORR) to pralatrexate treatment in Asian PTCL patients after prior treatment failure, as determined by independent imaging reviewer(s) using international workshop lymphoma response criteria (IWC)

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | Up to 40 weeks
  Incidence of adverse events (AE) and serious adverse events (SAE) emergent from the treatment
Overall survival | Up to 5 years
  Duration of overall survival (months)
Progression-free survival | Up to 5 years
  Duration of PFS (months)
Completion response rate | Up to 5 years
  The percentage of CR
Partial response rate | Up to 5 years
  The percentage of PR
Duration of CR and PR | Up to 5 years
  Duration of completion response and partial response (days)
Treatment duration | Up to 35 weeks
  Treatment duration with pralatrexate in the patients without HSCT who achieve CR or PR
Hematopoietic stem cell transplant (HSCT) | Up to 5 years
  Percentage of patients who undergo HSCT
1-year OS rate after HSCT | Up to 1 year
  1-year overall survival rate after conducting HSCT
1-year PFS rate after HSCT | Up to 1 year
  1-year progression-free survival rate after conducting HSCT
1-year relapse rate after HSCT | Up to 1 year
  1-year relapse rate after conducting HSCT
2-year OS rate after HSCT | Up to 2 years
  2-year overall survival rate after conducting HSCT
2-year PFS rate after HSCT | Up to 2 years
  2-year progression-free survival rate after conducting HSCT
2-year relapse rate after HSCT | Up to 2 years
  2-year relapse rate after conducting HSCT

CONTACTS AND LOCATIONS:
Overall Officials: Bor-Sheng Ko, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- Ntional Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Savage KJ. Peripheral T-cell lymphomas. Blood Rev. 2007 Jul;21(4):201-16. doi: 10.1016/j.blre.2007.03.001. Epub 2007 May 18. PMID 17512649
- [Background] Shustov A. Novel therapies for peripheral T-cell lymphomas. Ther Adv Hematol. 2013 Jun;4(3):173-87. doi: 10.1177/2040620713481980. PMID 23730495
- [Background] Savage KJ, Harris NL, Vose JM, Ullrich F, Jaffe ES, Connors JM, Rimsza L, Pileri SA, Chhanabhai M, Gascoyne RD, Armitage JO, Weisenburger DD; International Peripheral T-Cell Lymphoma Project. ALK- anaplastic large-cell lymphoma is clinically and immunophenotypically different from both ALK+ ALCL and peripheral T-cell lymphoma, not otherwise specified: report from the International Peripheral T-Cell Lymphoma Project. Blood. 2008 Jun 15;111(12):5496-504. doi: 10.1182/blood-2008-01-134270. Epub 2008 Apr 2. PMID 18385450
- [Background] Society TLL, Peripheral T-Cell Lymphoma Facts, 2014.
- [Background] Wang ES, O'Connor O, She Y, Zelenetz AD, Sirotnak FM, Moore MA. Activity of a novel anti-folate (PDX, 10-propargyl 10-deazaaminopterin) against human lymphoma is superior to methotrexate and correlates with tumor RFC-1 gene expression. Leuk Lymphoma. 2003 Jun;44(6):1027-35. doi: 10.1080/1042819031000077124. PMID 12854905
- [Background] Krug LM, Ng KK, Kris MG, Miller VA, Tong W, Heelan RT, Leon L, Leung D, Kelly J, Grant SC, Sirotnak FM. Phase I and pharmacokinetic study of 10-propargyl-10-deazaaminopterin, a new antifolate. Clin Cancer Res. 2000 Sep;6(9):3493-8. PMID 10999734
- [Background] O'Connor OA, Pro B, Pinter-Brown L, Bartlett N, Popplewell L, Coiffier B, Lechowicz MJ, Savage KJ, Shustov AR, Gisselbrecht C, Jacobsen E, Zinzani PL, Furman R, Goy A, Haioun C, Crump M, Zain JM, Hsi E, Boyd A, Horwitz S. Pralatrexate in patients with relapsed or refractory peripheral T-cell lymphoma: results from the pivotal PROPEL study. J Clin Oncol. 2011 Mar 20;29(9):1182-9. doi: 10.1200/JCO.2010.29.9024. Epub 2011 Jan 18. PMID 21245435